CLINICAL TRIAL: NCT01542671
Title: Tailored Lifestyle Intervention in Obese Adults Within Primary Care Practice
Brief Title: Tailored Lifestyle Intervention in Obese Adults Within Primary Care Practice - Choose to Lose
Acronym: CTL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Hospital of Rhode Island (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Charles B. Eaton, Principal Investigator, Memorial Hospital of Rhode Island
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 09-32; 5R18DK079880 (NIH)
Record Dates: First submitted 2012-02-27; First posted 2012-03-02 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-03

CONDITIONS: Overweight and Obesity
Keywords: lifestyle change; obesity treatment; physical activity; primary care; quality of life
MeSH Terms: conditions — Overweight; Obesity; Motor Activity | interventions — Methods

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Lifestyle counseling at baseline, six, twelve months; Food and exercise log recording and feedback, motivational phone calls monthly for 12 months, 4 tailored mailings on lifestyle change, and weekly mailings on weight loss, exercise, and healthy eating for first 12 months. Maintenance mailings biweekly for six months and then monthly during the second year.
  Interventions: Behavioral: Intervention
- Control (Placebo Comparator): Lifestyle counseling at baseline, six and twelve months similar to intervention group, and infrequent non-tailored pamphlets.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Intervention — * Lifestyle Counselor meetings at baseline, 6 months, and 12 months
  * Structured eating plan
  * Tailored nutritional and exercise tips. Weekly: months 1-12, biweekly: months 13-18, and monthly: months 19-24.
  * Monthly Motivational phone calls with Lifestyle Counselor for the first year
  * 4 informational DVDs over the two year period
  * Feedback on submitted food and exercise journals
  Arms: Intervention
Behavioral: Control — * Lifestyle Counselor meetings at baseline, 6 months, and 12 months
  * Structured eating plan
  * 5 informational NIDDK mailings over the two year period
  Arms: Control

SUMMARY:
The primary objective of the study is to evaluate the effectiveness of tailored lifestyle intervention in primary care by comparing changes in the primary measure of weight and body mass index (BMI) and secondarily: physical activity (PA), fat calories consumed, and fruit/vegetable servings within the two arms (intervention and control) of the study. It is hypothesized that the intervention cohort will demonstrate greater reductions in body weight, body neglect, and fat calories consumed and greater increases in physical activity and fruits/vegetable servings after two years compared to the control cohort. The study also aims to evaluate and compare the cost of intervention for purpose per each unit of measure lost between the two arms of the study as a secondary objective. The cost of intervention will be evaluated as it relates to study replication.

DETAILED DESCRIPTION:
The study will translate and evaluate previously successful weight loss and physical activity studies into a primary care setting in terms of efficacy and cost effectiveness. Patients are recruited by their primary care physicians office and screened for participation and contraindications by phone. A screening visit with a run-in period of food and exercise log adherence is performed. All participants have meetings with a Lifestyle Counselor to set nutritional and lifestyle goals and an introduction to weight loss techniques at baseline, 6 months, and 12 months. A structured eating plan will be given at the baseline visit. Participants at the baseline visit are randomized to either the intervention and control groups. During the first year, intervention participants will receive monthly motivational phone calls from their lifestyle counselor to assess their progress and help navigate the lifestyle changes. Food and exercise logs are reviewed frequently and written feedback give to each interventional participant. Intervention participants also receive weekly mailings focusing on weight loss, physical activity and healthy eating, and four tailored mailings based upon information gained through contact with the lifestyle counselor. Intervention participants will also receive 2 informative DVDs during the first year. Control participants receive 2 NIDDK informational handouts on weight loss. For the second year of the study focuses on maintenance. Intervention participants receive reduced mailings of 2 per month for 6 months and then once a month until the end of one year. Intervention participants receive one additional motivational phone call at 13 months if they have not reached their weight loss goal and also receive 2 more informative DVDs. The control participants will receive 3 informational NIDDK mailings. The two arms of the study will be compared using the critical outcome measures (weight loss, PA, fat calories & vegetable/fruit servings consumed) and secondary outcome measures (waist and hip circumference,BP,Heart rate) for weight loss efficacy. We will also evaluate the cost-effectiveness for dissemination as a PCP weight loss program in addition to the overall cost-effectiveness for the participant in terms of money spent and adverse events related to the lifestyle change.

ELIGIBILITY:
Inclusion Criteria:

* Male/female ≥18 and <80 years old
* Available for this research project for the entire 24-month study period
* Able to read and speak English
* Can provide informed consent

Exclusion Criteria:

* Diagnosed or hospitalization for active CVD disease in the past 6 months including: CHD or history of coronary revascularization procedure (e.g. angioplasty, bypass graft surgery), Stroke, Peripheral Vascular Disease, Heart Failure, Deep Vein Thrombosis (DVT)
* Unstable psychiatric condition
* History of a significant orthopedic limitation or other conditions that make exercise dangerous or extremely difficult
* Limited physical activity by a physician to less than a brisk walk
* Another family member in the study
* Limited prescribed diet (e.g. gluten free diet)
* Present treatment for an eating disorder
* Underwent treatment for cancer in the past 5 years
* Dialysis
* Poorly controlled diabetes (HgbA1c > 10) or hospitalized in past 6 months for poorly controlled diabetes
* Chronic steroid therapy
* Participant requesting surgical treatment of obesity or weighing over 400 lbs.
* Major surgery in the past month
* Participating in another clinical trial with regards to obesity or physical activity

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2009-09; Primary Completion 2014-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Changes in Body Weight & Physical Activity | Five years
  The primary outcomes of the trial are measured changes in BMI and physical activity level.

SECONDARY OUTCOMES:
Cost Effectiveness | Five Years
  Secondary outcomes are cost effectiveness of the intervention as measured by cost per unit of BMI loss. Additional outcomes are changes in stages of change, decision balance, self-efficacy, and problem solving skills during the trial.
Eating Behaviors | 5 years
  Eating behaviors (measured as servings of fruits/vegtables and fat calories consumed) as self reported, Diet History Questionnaire II, SF-12, Eating Behavior Inventory, Three Factor Eating, and General Self Efficacy questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Charles B Eaton, MD, Principal Investigator — Memorial Hospital of Rhode Island
Locations (1):
- Memorial Hospital of Rhode Island, Pawtucket, Rhode Island, United States